CLINICAL TRIAL: NCT03408106
Title: Prospective Clinical Trial of HIV+ Living Donor Kidney Donation for HIV+ Recipients
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00138153
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective Clinical Trial of HIV+ Living Donor Kidney Donation for HIV+ Recipients

DETAILED DESCRIPTION:
This is a prospective study to evaluate the safety of donor nephrectomy in HIV+ individuals who donate kidneys to HIV+ candidates in need of transplant . The study will assess potential complications of HIV + living donors - including adverse events related to nephrectomy, development of chronic kidney disease, hypertension, and HIV-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide consent
* Age 21 years or older
* Meets standard clinical criteria for living donation per Johns Hopkins University (JHU) Comprehensive Transplant Center Policy
* Documented HIV infection (by any licensed Enzyme-linked Immunosorbent Assay (ELISA) and confirmation by Western Blot, positive HIV Ab Immunofluorescent Assay (IFA), or documented history of detectable HIV-1 RNA)
* CD4+ T-cell count ≥ 500/µL for 6 months prior to donation
* HIV-1 RNA below 50 copies RNA/mL (viral blips between 50-400 copies will be allowed as long as there are not consecutive measurements >200 copies/mL)

Exclusion Criteria:

* Two high risk alleles of APOL1 (G1 or G2 variants)
* Hypertension
* Diabetes
* Chronic active hepatitis C (detectable HCV RNA in plasma)
* Evidence of invasive opportunistic complications from HIV infection
* Mentally incompetent and/or inability to provide informed consent
* Other medical conditions, as determined by the provider, that would preclude donation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV+ patients 21 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | at 1 year
  incidence of adverse events related to nephrectomy

SECONDARY OUTCOMES:
chronic kidney disease | through to study completion, up to 4 years
  time to significant proteinuria or glomerular filtration rate below 60 ml/min
hypertension | through to study completion, up to 4 years
  time to hypertension defined as systolic blood pressure > 140 mm Hg confirmed
change in antiretroviral therapy | through to study completion, up to 4 years
  proportion of participants requiring change in antiretroviral therapy
HIV virologic control | through to study completion, up to 4 years
  proportion of participants with HIV virologic failure or breakthrough

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland